CLINICAL TRIAL: NCT05351294
Title: Assessment of Early Radiation Oncology Involvement Alongside Standard Oncologic Care in the Management of Metastatic Malignancies
Brief Title: Assessment of Early Radiation Oncology Involvement Alongside Standard Oncologic Care in the Managemet
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Malcolm David Mattes, MD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002168; Pro2021002435 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-03-15; First posted 2022-04-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Radiation Therapy; Metastatic Cancer
Keywords: Quality of Life; Palliative Care and Supportive Care
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): All enrolled patients will receive standard oncologic care at the discretion of the treating physicians, but will also complete the EORTC QLQ-C30, EQ-5D-5L, PTPQ, FAMCARE-P16 at baseline before randomization. Follow-up assessment using EORTC QLQ-C30, PTPQ, FAMCARE-P16 will occur every 3 months, and using EQ-5D-5L will occur every 1 month, for a total of 12 months. These will be administered during standard-of-care clinic or infusion center visits.
  Interventions: Other: Questionnaires
- Arm 2 (Experimental): Patients enrolled in Arm 2 will also be seen be a radiation oncologist during the course of the study. The RO will review the patient's most recently completed EQ 5D-5L questionnaires and perform a complete History and Physical evaluation to determine if there is any immediate role for PRT. Based on the patient's type of cancer and areas of spread, the RO will also discuss types of symptoms that could develop in the future, and give instructions and educational materials to the patient so he/she can better identify those symptoms early on.
  Interventions: Combination Product: Early Radiation Oncology Involvement Alongside Standard Oncologic Care

INTERVENTIONS:
Other: Questionnaires — All patients in Arm 2 will be seen and treated by one of three ROs with an interest in participating in this study, who will be trained by the PI to perform these visits reproducibly and with rigor. These will all be "regular" ROs, who like most ROs administer a mix of curative and PRT in their clinical practice; like most cancer centers, there are no ROs who formally subspecialize in PRT at our institution. Notably, patients in Arm 1 (control arm) will always have standard-of-care RO referral available for consideration of PRT if needed for symptom relief. However, patients in Arm 1 will be seen by other ROs without any specific training for this study. Any courses of PRT administered in either arm are at the discretion of the treating RO in terms of the timing, dose, fractionation, and treatment technique.
  Arms: Arm 1
Combination Product: Early Radiation Oncology Involvement Alongside Standard Oncologic Care — Early Radiation Oncology Involvement Alongside Standard Oncologic Care
  Arms: Arm 2

SUMMARY:
To determine if the experimental approach of early radiation oncology involvement alongside standard oncologic care will result in higher HRQL at 6 months compared to the control arm receiving standard oncologic care alone, based on the global subscale score of the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire.

DETAILED DESCRIPTION:
Primary Objective To determine if the experimental approach of early radiation oncology involvement alongside standard oncologic care will result in higher HRQL at 6 months compared to the control arm receiving standard oncologic care alone, based on the global subscale score of the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire. Secondary Objectives

1. To determine if early radiation oncology involvement improves other more detailed metrics of HRQL. This will be assessed using each of the 5 domains of the EORTC QLQ-C30 (physical, role, cognitive, emotional, social), each of the 5 dimensions of the EuroQol (EQ) 5D-5L (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), and the health index score and EQ visual analogue scale. If there are significant differences in the primary endpoint, then a cost-utility analysis will be conducted using a Markov model and the EQ-5D-5L index scores.
2. To determine if early radiation oncology involvement will reduce the incidence of severe exacerbations/crises in cancer-induced symptoms (excluding systemic therapy-induced side effects), according to the number of emergency department visits and hospitalizations (total number of occurrences, and days admitted). These findings will be reported in the context of the number of palliative radiation therapy (PRT) courses and other invasive procedures that patients undergo, toxicities from those treatments, duration of time to initiation of tumor-directed treatment for exacerbation in symptoms, number of different lines of systemic therapy administered, and overall survival of each patient.
3. To determine if early radiation oncology involvement improves other metrics of quality palliative care across the disease trajectory, as assessed by rates of early Palliative and Supportive Care (PSC) referral alongside standard oncologic care, documented advance care planning (based on the percentage of patients in both arms who complete a living will, and designate a power of attorney and resuscitation preferences in the medical record), hospice referral prior to death, and aggressiveness of care within 14 days of death (defined as meetings any of the following three criteria: chemotherapy, radiation, or surgery within 14 days before death, no hospice care, or admission to hospice 3 days or fewer before death).
4. To assess patient/caregiver perceptions of prognosis, goals of treatment, and quality of communication with oncologists through the use of the Prognosis and Treatment Perceptions Questionnaire (PTPQ) in each arm
5. To assess satisfaction with information-giving, availability of care, psychological care, and physical care in patients with advanced cancer using the FAMCAREP16 questionnaire in each arm
6. To assess caregiver burden using the Montgomery-Borgatta Caregiver Burden Scale.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for this study are as follows:

1. Age ≥ 18 years
2. Zubrod performance status 0-2
3. Pathology-proven cancer, with primary site outside of the central nervous system
4. Clinical (based on physical exam or imaging) or pathological diagnosis of metastatic disease, for which curative intent treatment is not feasible and treatment goals are palliative. Both patients with newly diagnosed metastatic disease, and those who have a metastatic relapse after prior curative-intent treatment for their malignancy, are eligible.
5. Estimated life expectancy 6-24 months. Guidelines for estimating life expectancy will be based on best available evidence, based primarily on tumor type, systemic therapy used and its expected outcome, line of systemic therapy, and in some cases patients' initial response to systemic therapy, along with the enrolling medical oncologist's judgement.
6. Either planned, or actively receiving, systemic therapy (chemotherapy, targeted/biologic therapy, immunotherapy, or hormonal therapy)
7. Ability to understand and the willingness to sign a written informed consent document
8. If a patient is actively participating in another clinical trial utilizing an investigation agent, they are still eligible for participation in this study unless radiation therapy is explicitly not allowed in that trial.

Exclusion Criteria:

The exclusion criteria for this study are as follows:

1. Patients with metastatic solid tumors but life expectancy longer than 24 months will be excluded. This list includes (but is not limited to):

   1. Castrate-sensitive prostate cancer (castrate-resistant prostate cancer are eligible)
   2. Breast cancer responsive to hormonal therapy
   3. Endometrial cancer responsive to hormonal therapy
   4. Patients receiving first line systemic therapy, for whom median progression-free survival is greater than 6 months, and response to therapy has not been assessed yet.
2. Patients considered metastatic only due to pleural or peritoneal metastases without metastases to any other organ are excluded since palliative radiation therapy is less commonly used in these cases.
3. Patients with cancer considered incurable that is locally advanced but nonmetastatic.
4. Patients with leukemia or primary central nervous system cancers will be excluded since these patients less commonly are treated with palliative radiation therapy. Patients with lymphoma and multiple myeloma are eligible if they meet the other eligibility criteria.
5. Any patient for whom standard-of-care radiation oncology referral would be immediately indicated for palliative radiation therapy. The purpose of this is to ensure that patients in the control arm will not have a detriment in their care by not seeing a radiation oncologist at enrollment,
6. In order to avoid bias from prior standard-of-care radiation oncology involvement, patients will also be excluded if they are undergoing active follow-up with a radiation oncologist after prior palliative radiation therapy.
7. History of whole brain radiation therapy for brain metastases (patients who underwent one prior treatment with radiosurgery for brain metastases are eligible)
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, adrenal insufficiency, chronic liver disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Pregnant or breastfeeding women; Subjects who are pregnant are excluded from this study because radiation therapy has the potential for teratogenic or abortifacient effects.
10. Cognitively impaired adults lacking decision-making capacity or unable to consent. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Measure of Health-related quality of life (HRQL) at six months | At Six Months
  To see if early radiation oncology involvement alongside standard oncologic care will result in higher Health-related quality of life (HRQL) at six months compared to the control arm receiving standard oncologic care alone, based on the global subscale score of the European Organization for Research and Treatment of Cancer(EORTC) QLQ-C30 questionnaire.

SECONDARY OUTCOMES:
Levels of HRQL | 12 Months
  To measure health-related quality of life (HRQL), by seeing if early radiation oncology involvement improves other more detailed metrics of HRQL.
Health Index Score | 12 months
  To measure the degree of severity or damage incurred by an organ or tissue.

OTHER OUTCOMES:
Vertical Visual Analogue Scale (EQ visual analogue scale) | 12 months
  Participants will measure the assessment of their health
EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) | 12 months
  To measure cancer participants physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Mattes, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (6):
- United States (6):
  - RWJBarnabas Health Jersey City Medical Center, Jersey City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Malcolm David Mattes, MD, Newark, New Jersey
  - RWJBarnabas Health - Newark Beth Israel Medical Center, Newark, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Somerset, New Jersey

IPD SHARING:
Plan to Share IPD: No